CLINICAL TRIAL: NCT01861652
Title: The Use of the Vasculaire Leg Compression Device for the Treatment of Restless Legs Syndrome - A Prospective Clinical Study
Brief Title: Vasculaire Leg Compression Device for the Treatment of Restless Legs Syndrome - A Prospective Clinical Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor withdrew support
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 388140
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2013-05

CONDITIONS: Restless Legs Syndrome,; Restless Legs,; Ekbom Syndrome
Keywords: Restless legs syndrome, Ekbom syndrome, Restless legs
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Venous health systems Vasculaire leg compression device (Experimental): Vasculaire leg compression device
  Interventions: Device: Venous Health Systems Vasculaire Leg Compression Device

INTERVENTIONS:
Device: Venous Health Systems Vasculaire Leg Compression Device — Leg (calf) compression device used to alleviate symptoms of restless legs
  Other Names: intermittent pneumatic compression device; sequential intermittent pneumatic compression device

SUMMARY:
Restless legs syndrome (RLS) is a debilitating sleep disorder that has significant impact on quality of life, and often times can be difficult to diagnose and treat effectively. RLS is typically treated with medical therapy (including dopaminergic agents, dopamine agonists, benzodiazepines, anticonvulsants, opiates, among other therapies). Many patients are either refractory to medical therapy, have contraindications or adverse reactions to the available medical therapies, or desire conservative non-medication based therapies. Two previous studies have demonstrated that pneumatic compression devices placed on the legs can improve symptoms of RLS. We would like to assess whether the Venous Health Systems Vasculaire leg compression device improves symptoms and quality of life measures related to RLS in up to 40 patients evaluated prospectively for one month. This is a pilot study to assess the subjective response of our cohort of patients to this device prospectively. Our hypothesis is that over 66% of our cohort will demonstrate a positive symptomatic response based on RLS specific quality of life questionnaires.

DETAILED DESCRIPTION:
BACKGROUND:

Restless Leg Syndrome (RLS) affects nearly 12 million Americans. Although the precise etiology of RLS is not well characterized, there are specific diagnostic criteria. Symptoms are typically worse in the evening, consisting of a strong urge to move the affected limb(s) and relief with movement. Current medical therapies pose several challenges for many patients, as side effects include extreme drowsiness, hallucinations, nausea, headaches and insomnia. An alternative, non-medical therapy may provide a suitable option to this subset of patients. Intermittent pneumatic compression devices have previously been studied in this population, and have demonstrated effectiveness. However prior models have required subjects to remain immobile during use, representing a significant limitation given that immobility may actually promote worsening of symptoms. An effective, alternative non-pharmacologic therapy that does not interfere with patient mobility should provide a valuable treatment option.

The purpose of this study is to assess whether the Vasculaire Intermittent Pneumatic Compression System will improve validated measures of symptom relief, patient satisfaction, and quality of life for RLS. This is a pilot study to determine whether or not the Vasculaire device improves validated measures of symptom relief, patient satisfaction, and quality of life in RLS patients. Depending on the outcome of our study we hope to develop a sham-controlled clinical trial as a follow-up study.

METHODS:

We are performing a Prospective cohort study.

We will recruit patients until we reach an N=40.

After informed consent, the patient's record will be reviewed to ensure that they have had a serum iron panel and ferritin checked within the preceding 6 months. For those patients missing these laboratory studies, they will have their blood drawn for a full serum iron panel (serum iron level, serum ferritin, and total iron binding capacity), as per standard of care (to exclude iron deficiency as a cause or contributor to their symptoms). Patients with inadequate serum iron stores will be excluded. Patients with adequate iron stores will be asked to complete a comprehensive medical questionnaire to document medical conditions and medications with doses prescribed.

This questionnaire will also record previously tried therapies, both home remedies and medically prescribed treatments. Specific undesirable side effects will also be documented.

Severity will then be determined based on 5 previously validated questionnaire instruments (The Restless Legs Syndrome Rating Scale, The Restless Legs Syndrome-Quality of Life Instrument (RLS-QLI), The Epworth Sleepiness Scale (ESS), The Johns Hopkins Restless Legs Severity Scale (JHRLS), The International Restless Legs Syndrome Rating Scale).

Once the medical history has been reviewed, documentation of severity assessed and the determination of unresolved treatment post medical therapy, the patient will be eligible for enrollment.

The Vasculaire Intermittent Pneumatic Compression System will be introduced to the patient and instructions provided on how to optimize the use of device in accordance with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are at least 18 years of age with a reliable diagnosis of RLS in accordance with the International Classification of Sleep Disorder, Revised Diagnostic and Coding Manual of the American Academy of Sleep Medicine. All patients included must have persistent symptoms that interfere with quality of life. Patients who are currently on approved medical therapy for RLS must be on a stable dose/agent for ≥30 days and experience persistent symptoms that interfere with quality of life. Patients who are currently refractory to medical therapies may also be included if they are presently under the care of a physician and receiving medical therapy for RLS for ≥30 days without improvement and/or having experienced unacceptable side effects. Pregnancy status is not being assessed and is not relevant to device use.

Exclusion Criteria:

* Younger than 18 years, unstable medical conditions that may interfere with the requirements of the study, e.g. diabetes mellitus, symptomatic asthma, congestive heart failure with nocturnal symptoms, and mental or physical limitation (including dementia) that would preclude data collection on questionnaires or wearing intermittent pneumatic compression devices. Other medical conditions that would serve as exclusion criteria are those where increased venous or lymphatic return is undesirable. These specific conditions are known or suspected deep vein thrombosis, thrombophlebitis, severe congestive heart failure, pulmonary edema, severe arteriosclerosis, action infection such as gangrene, recent vein ligation or skin graft, or extreme deformity of the legs. Patients with iron deficiency anemia, or evidence of inadequate serum iron stores on laboratory testing are also excluded until this has been corrected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The Restless Legs Syndrome Rating Scale | one month
  the patient rates their symptoms of RLS on a severity scale (none (0), mild (1-10), moderate (11-20), severe (21-30), very severe (31-40))
The Restless Legs Syndrome-Quality of Life Instrument (RLS-QLI) | one month
  18 questions assessing how RLS has affected patient's quality of life over the preceding month.
The Epworth Sleepiness Scale (ESS) | one month
  A validated questionnaire for assessing daytime sleepiness; propensity to fall asleep during routine daily tasks/events.
The Johns Hopkins Restless Legs Severity Scale (JHRLS) | one month
  assesses how severe a patient's RLS symptoms are at different points in the day (symptoms occuring earlier in the day is worse). Severity graded as 0=never, 0.5=infrequent, 1=mild, 2=moderate, 3=severe, 4=very severe
The International Restless Legs Syndrome Rating Scale | 1, 2, 3, 4 weeks
  assesses a patient's symptoms of RLS over the preceding week in terms of severity (numeric score)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob F Collen, MD, Principal Investigator — Pulmonary, Critical Care, Sleep Medicine; Christopher J Lettieri, MD, Study Director — Pulmonary, Critical Care, Sleep Medicine
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lettieri CJ, Eliasson AH. Pneumatic compression devices are an effective therapy for restless legs syndrome: a prospective, randomized, double-blinded, sham-controlled trial. Chest. 2009 Jan;135(1):74-80. doi: 10.1378/chest.08-1665. Epub 2008 Nov 18. PMID 19017878
- [Background] Eliasson AH, Lettieri CJ. Sequential compression devices for treatment of restless legs syndrome. Medicine (Baltimore). 2007 Nov;86(6):317-323. doi: 10.1097/MD.0b013e31815b1319. PMID 18004176